CLINICAL TRIAL: NCT05337540
Title: A Double-Blind, Randomized, Controlled, Three Parallel Arm, Dose-Finding Study to Evaluate the Efficacy, Safety and Tolerability of One Single Intra-Articular Injection of EVI-01 in Patients With Symptomatic Osteoarthritis of the Knee
Brief Title: A Study to Evaluate the Efficacy, Safety and Tolerability of EVI-01 Intra-Articular Injection in Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aptissen SA (Industry)
Collaborators: Azidus Brasil (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EVI-01-BR
Record Dates: First submitted 2022-04-14; First posted 2022-04-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EVI-01 - low dose (Experimental): 4 mL, one single EVI-01 intra-articular injection
  Interventions: Device: EVI-01
- EVI-01 - high dose (Experimental): 6 mL, one single EVI-01 intra-articular injection
  Interventions: Device: EVI-01
- Synvisc-One (Active Comparator): 6 mL, one single intra-articular injection
  Interventions: Device: Active comparator Synvisc-One

INTERVENTIONS:
Device: EVI-01 — Single intra-articular injection of high molecular weight hyaluronic acid
  Arms: EVI-01 - high dose; EVI-01 - low dose
Device: Active comparator Synvisc-One — Single intra-articular injection of active comparator Synvisc-One
  Arms: Synvisc-One

SUMMARY:
Objective: Identifying the dose of EVI-01 with the best clinical response, balancing the efficacy, safety, and tolerability of the investigational product.

Study design: Interventional, dose-finding, three arms, randomized (1:1:1), parallel assignment, double-blind, controlled by an active comparator.

DETAILED DESCRIPTION:
Phase II, dose-finding, interventional, three-arm, randomized (1:1:1), double-blind, parallel, active-comparator-controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders aged 18 years or older;
2. Body Mass Index (BMI) < 35 kg/m2;
3. Diagnosis of primary knee osteoarthritis, Kellgren-Lawrence Grade 2 to 4, according to American College of Rheumatology (ACR) criteria and confirmed radiologically within the previous 12 months, for which an intraarticular treatment is indicated;
4. Moderate to severe pain measured by VAS (0-100mm) and >40mm in the knee to be treated, partially responsive to chronic doses of nonsteroidal anti-inflammatory drugs (NSAIDs), analgesics, or weak opioids (codeine and tramadol);
5. Ability to understand and provide signed consent through the Informed Consent Form (ICF).

Exclusion Criteria:

1. History of hypersensitivity/allergy to hyaluronic acid (HA) or other excipients of the IP or product;
2. Pregnant or breastfeeding women;
3. Women at menace who do not agree to use acceptable contraceptive methods (oral contraceptive, injectable contraceptive, IUD, hormonal implant, barrier methods, sexual abstinence, hormone transdermal patch and tubal ligation); except those who are surgically sterile (bilateral oophorectomy or hysterectomy);
4. Emotional problems or any situation that, at the Investigator's discretion, places the safety of subjects at risk;
5. Application of visco-supplementation to the knee less than four months prior to randomization;
6. Corticosteroid IA injection less than 4 months prior to randomization and/or schedule during the course of the study;
7. Knee infection and/or inflammation (e.g., bursitis), skin infection at or around the IA injection;
8. Swelling, redness, warmth, or other clinically relevant inflammatory signs in the knee in the investigator's description
9. Knee injury or trauma;
10. Patients with bleeding diathesis or on anticoagulant therapy;
11. Major knee malformations or deformities that the investigator deems pertinent;
12. Active cancer at the Investigator's discretion;
13. Continuous or frequent use (use for more than 2 weeks in the last 2 months) of corticosteroids by any route of administration (oral, IM, IV)
14. Concomitant use of chondroprotective drugs such as glucosamine, chondroitin, or collagen. These medications should not be introduced during the study, but if the patient is already taking them may be included, but the medication will not change.
15. Need for the use of strong opioids (methadone, fentanyl, morphine, and oxycodone) for pain management;
16. Participation in a clinical trial within the last twelve months prior to enrollment (CNS Resolution 251, dated 07 August 1997, item III, item J), unless the investigator believes that there may be a benefit to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Changes to the questionnaire WOMAC A (Western Ontario and McMaster Universities) Numeric 3.1 | from baseline to 180 days after randomization
  Questionnaire WOMAC A (Western Ontario and McMaster Universities) numeric scale, version 3.1, total knee pain score (pain, stiffness and physical function assessment)
Comparison of treatment-related Adverse Events in the three groups | from baseline to 180 days after randomization
  Incidence of treatment-emergent adverse events

SECONDARY OUTCOMES:
Changes to the WOMAC (Western Ontario and McMaster Universities) Total Numeric 3.1 score | from baseline to 180 days after randomization
  WOMAC (Western Ontario and McMaster Universities) numeric scale, version 3.1 (pain, stiffness and physical function assessment)
Changes to the WOMAC (Western Ontario and McMaster Universities) A score | from Day 1 to Day 7 after randomization
  WOMAC (Western Ontario and McMaster Universities) A numeric scale, version 3.1, total knee pain score (pain, stiffness and physical function assessment)
Response to the Euro Quality of Life Questionnaire | from baseline to 180 days after randomization
  Euro Quality of Life Questionnaire version EQ-5D-5L
Response rate, according to OMERACT-OARSI2 international criteria | from baseline to Days 28, 90 and 180 after randomization
  OMERACT-OARSI2 (Outcome Measures in Rheumatology Committee - Osteoarthritis Research Society International)

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Gracitelli, MD, Principal Investigator — C.E.P.O.T. - Centro de Estudos e Pesquisas em Ortopedia e Traumatologia
Locations (2):
- Brazil (2):
  - A2Z Clinical, Valinhos, São Paulo
  - Ortocity, São Paulo